CLINICAL TRIAL: NCT05855096
Title: Clinical Assessment And Treatment Preferences of Physiotherapists Working in Neurorehabilitation: A Research From Turkey
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Other Study IDs: Biruni Un
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Neurorehabilitation; Physiotherapist; Clinical Assessment; Treatment Preferences
Keywords: neurorehabilitation; physiotherapist; perspectives

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Google Form Questionnaire — Google form questionnaire is performed by responders.

SUMMARY:
The most common neurological diseases are stroke, Multiple Sclerosis and Parkinson's. Neurorehabilitation is a process that aims to improve the quality of life by minimizing the functional disorders caused by the motor and sensory effects of the problems in the nervous system. A detailed and accurate evaluation and an effective treatment program are required for successful neurorehabilitation. There is no common perspective on evaluation and treatment methods used in the field of neurorehabilitation.The aim of this study is to establish a standard perspective by determining the most preferred evaluation and treatment methods by physiotherapists working in the field of neurorehabilitation in our country. This perspective will help to establish a common understanding in the field of neurorehabilitation and to have knowledge of the different methods used by all physiotherapists working in this field. In this way, the treatment process of the patients will become more effective, and the results obtained from the treatment will be reflected positively. This study will be a resource showing the evaluation methods and preferences of physiotherapists working in the field of neurorehabilitation in Turkey.

DETAILED DESCRIPTION:
Rehabilitation is a part of health services performed in many diseases and specific areas. It has four stages, and these are prevention, enhancement, treatment and protection. The main purpose of rehabilitation programs is independence in activities. It is to increase the quality of life and social adaptation of the patient by protecting the patient, minimizing pain and disability, and improving the ability to adapt to changing conditions. Neurological problems are one of the areas that often need rehabilitation. Millions of people worldwide are affected by neurodegenerative problems. According to the data shared by the World Health Organization (WHO), many of the neurological disorders are chronic and progressive, creating a global picture. Neurological problems negatively affect the health of the individual in many ways. To improve the physical and emotional functions, quality of life and social participation levels of individuals with neurological disease, it is necessary to know the limitations they experience due to neurological disease very well. The causes of neurological problems can vary from person to person and from problem to problem. These causes may include genetic disorders, congenital abnormalities or disorders, infections, lifestyle, or environmental health issues, including malnutrition, brain injury, spinal cord injury, nerve injury [8,9]. In addition, the neurological problem may begin in another system that interacts with the nervous system. For example, stroke (cerebrovascular accident), includes brain damage caused by problems with the blood vessels that feed the brain (cardiovascular system); autoimmune disorders, caused by the body's own immune system includes damage. Neurological diseases bring with them secondary problems besides primary problems. These secondary problems and deformities negatively affecting function, productivity and participation, which are essential components of their activities, restricts the independence of the individual. Pertaining to the motor and sensory systems seen in neurological diseases. The problems are often accompanied by cognitive, behavioural, sensory, communication and perception disorders. is seen. It is known that participation in daily life activities is one of the elements that increase the creativity of individuals, improve their skills and enable them to integrate into social life .By identifying the limitations experienced by individuals due to neurological disease. Improving their quality of life and social participation levels is the most basic of rehabilitation is the target. The most common neurological diseases are stroke, Multiple Sclerosis and Parkinson's. Neurorehabilitation is a process that aims to improve the quality of life by minimizing the functional disorders caused by the motor and sensory effects of the problems in the nervous system. A detailed and accurate evaluation and an effective treatment program are required for successful neurorehabilitation.There is no common perspective on evaluation and treatment methods used in the field of neurorehabilitation.The purpose of this study is to establish a standard perspective by determining the most preferred evaluation and treatment methods by physiotherapists working in the field of neurorehabilitation in our country. This perspective will help to establish a common understanding in the field of neurorehabilitation and to have knowledge of the different methods used by all physiotherapists working in this field. In this way, the treatment process of the patients will become more effective, and the results obtained from the treatment will be reflected positively. This study will be a resource showing the evaluation methods and preferences of physiotherapists working in the field of neuro rehabilitation in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Having at least 3 years of patient follow-up experience in the field of neurorehabilitation
* Men and women of all age groups who are in the active working process physiotherapists
* Being a volunteer
* Speaks and understands the Turkish language (for foreign nationals)

Exclusion Criteria:

* Respondents who did not or incompletely answered parts of the survey

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapists who can read and understand Turkish and have at least three years of work experience will be included in the study. It is planned to send the questionnaire prepared via Google Survey to physiotherapists working in the field via non-governmental organizations, social media and association mails. In the questionnaire, it was aimed to question the age, gender, duration of work in the profession, the duration of work in the field of neurorehabilitation, the training received after graduation, the most preferred evaluation and treatment methods for neurological diseases that are mostly encountered in the field.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Google Form Questionnaire | 5 minutes
  It is planned to send the questionnaire prepared via Google Questionnaire to the physiotherapists who accept to participate in the research and meet the inclusion criteria, to the physiotherapists working in the field via social media, the Physiotherapists Association of Turkey and its sub-groups registered members after the necessary permissions are obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Guzin Kaya Aytutuldu, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krug E, Cieza A. Strengthening Health Systems to Provide Rehabilitation Services. Ann Rehabil Med. 2017 Apr;41(2):169-170. doi: 10.5535/arm.2017.41.2.169. Epub 2017 Apr 27. No abstract available. PMID 28503447
- [Background] Wade DT. What is rehabilitation? An empirical investigation leading to an evidence-based description. Clin Rehabil. 2020 May;34(5):571-583. doi: 10.1177/0269215520905112. Epub 2020 Feb 10. PMID 32037876
- [Background] Guerra-Vazquez CM, Martinez-Avila M, Guajardo-Flores D, Antunes-Ricardo M. Punicic Acid and Its Role in the Prevention of Neurological Disorders: A Review. Foods. 2022 Jan 18;11(3):252. doi: 10.3390/foods11030252. PMID 35159404
- [Background] Ona ED, Cano-de la Cuerda R, Sanchez-Herrera P, Balaguer C, Jardon A. A Review of Robotics in Neurorehabilitation: Towards an Automated Process for Upper Limb. J Healthc Eng. 2018 Apr 1;2018:9758939. doi: 10.1155/2018/9758939. eCollection 2018. PMID 29707189
- [Background] Lexell J, Brogardh C. The use of ICF in the neurorehabilitation process. NeuroRehabilitation. 2015;36(1):5-9. doi: 10.3233/NRE-141184. PMID 25547759
- [Background] Zis P, Hadjivassiliou M. Treatment of Neurological Manifestations of Gluten Sensitivity and Coeliac Disease. Curr Treat Options Neurol. 2019 Feb 26;21(3):10. doi: 10.1007/s11940-019-0552-7. PMID 30806821
- [Background] Sanders T, Liu Y, Buchner V, Tchounwou PB. Neurotoxic effects and biomarkers of lead exposure: a review. Rev Environ Health. 2009 Jan-Mar;24(1):15-45. doi: 10.1515/reveh.2009.24.1.15. PMID 19476290
- [Background] McDowell FH. Neurorehabilitation. West J Med. 1994 Sep;161(3):323-7. No abstract available. PMID 7975575
- [Background] Tempest S, Jefferson R. Engaging with clinicians to implement and evaluate the ICF in neurorehabilitation practice. NeuroRehabilitation. 2015;36(1):11-5. doi: 10.3233/NRE-141185. PMID 25547760
- [Background] Krucoff MO, Rahimpour S, Slutzky MW, Edgerton VR, Turner DA. Enhancing Nervous System Recovery through Neurobiologics, Neural Interface Training, and Neurorehabilitation. Front Neurosci. 2016 Dec 27;10:584. doi: 10.3389/fnins.2016.00584. eCollection 2016. PMID 28082858
- [Background] van den Broek MD. Why does neurorehabilitation fail? J Head Trauma Rehabil. 2005 Sep-Oct;20(5):464-73. doi: 10.1097/00001199-200509000-00007. PMID 16170254